CLINICAL TRIAL: NCT06763705
Title: Evaluation of Safety and Efficacy of Non-anesthesia Provider-administered Different Anesthetic Regimens During Colonoscopy. Asingle Center, Prospective Double Blind, Randomized Study
Brief Title: Comparison of Safety and Efficacy for Different Sedation Regimens During Colonoscopy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Qassim Health Cluster (Other)
Responsible Party: Principal Investigator, Mohammed Saud Alsulaimi, Consultant gastroenterology, Qassim Health Cluster
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 607/45/15284
Record Dates: First submitted 2024-12-10; First posted 2025-01-08 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Deep Sedations; Conscious Sedation; Colonoscopy
Keywords: colonoscopy
MeSH Terms: interventions — Midazolam; Propofol; Fentanyl

STUDY DESIGN:
Intervention Model Description: a randomized, double-blinded study 3 arms study
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Midazolam + Fentanyl (Experimental): Midazolam AND Fentanyl Before start of colonoscopy procedure patient will be sedated with these drugs in this group. Doses: Midazolam: Initial dose 0.5-1 mg. Additional doses: 1 mg every 2-3 min depending sedation level, maximum dose: 6 mg. till completion of the colonoscopy procedure Fentanyl Initial dose: 12.5-75 μg Additional doses: 12.5-50 μg every 2-3 minutes. Maximum dose: 100 ug
  Interventions: Drug: Midazolam; Drug: Fentanyl
- Propofol (Experimental): Propofol Before start of colonoscopy procedure patient will be sedated with propofol in this group. Dose:induction dose of 20-50 mg followed by intermittent boluses of 10-20 mg according to the patient response. Maximum total dose of 200 mg. Till completion of the colonoscopy
  Interventions: Drug: Propofol
- Propofol +Fentanyl (Experimental): Propofol AND Fentanyl Before start of colonoscopy procedure patient will be sedated with these drugs in this group. Doses: Propofol: Induction dose of 20-50 mg followed by intermittent boluses of 10-20 mg according to the patient response. maximum total dose of 200 mg. Till completion of the colonoscopy procedure.
  Fentanyl Initial dose: 12.5-75 μg Additional doses: 12.5-50 μg every 2-3 minutes. Maximum dose: 100 ug. Till completion of the colonoscopy procedure
  Interventions: Drug: Propofol; Drug: Fentanyl

INTERVENTIONS:
Drug: Midazolam — It will not be used alone but in combination with Fentanyl in the Midazolam + Fentanyl group.
  Arms: Midazolam + Fentanyl
Drug: Propofol — It will used alone in Propofol group and in combination with Fentanyl in the Propofol + Fentanyl group.
  Arms: Propofol; Propofol +Fentanyl
Drug: Fentanyl — Fentanyl will not be used in isolation but will be used in combination with either Midazolam or Propofol in Midazolam + Fentanyl group and Propofol + Fentanyl group, respectively.
  Arms: Midazolam + Fentanyl; Propofol +Fentanyl

SUMMARY:
This is a randomized, double-blinded, prospective study which will be conducted at the Department of Gastroenterology, King Saud Hospital, Unaizah, Qassim, Saudi Arabia. This study aims to compare safety and efficacy of different types of sedation medications for elective colonoscopy. Colonoscopy is a procedure to examine and visualize the colon by a fiberoptic tube called colonoscope. Sedation helps one to relax to avoid feel any discomfort or pain during the procedure.

DETAILED DESCRIPTION:
The study will involve 157 patients who meet the inclusion criteria and are scheduled for elective colonoscopy. Sample size is calculated by ANOVA F test. Participants will be randomly assigned into three groups using computer-based randomization. Group I will receive intravenous midazolam + fentanyl, Group II will receive propofol only, and Group III will receive fentanyl + propofol. Dosages will be titrated as needed during the procedure, with sedation administered by trained nurses/doctors under the supervision of an anesthesiologist to ensure patient safety. Experienced endoscopists will perform the procedures, and all participants will undergo a pre-procedure evaluation, including medical history, physical examination, and assessment of allergies, comorbidities, and ASA classification. Data on patient demographics, procedure details, and sedative dosages will be collected, alongside monitoring of vital signs, oxygen saturation, and blood pressure before, during, and after the procedure.

The primary outcomes for the study include the degree of sedation, onset of sedation, patient satisfaction, and procedure completion rate. The degree of sedation will be assessed using the Observer's Assessment of Alertness/Sedation (OAA/S) scale, while the onset of sedation will be defined as the time it takes for the patient to show drowsiness and reduced responsiveness. Secondary outcomes include adverse events, recovery time, and endoscopist satisfaction. Adverse events, such as hypotension, tachycardia, bradycardia, and hypoxia, will be recorded using pre-defined criteria for each. Recovery will be assessed every 10 minutes post-procedure using the Aldrete score, with a score of 10 indicating full recovery, after which patients can be discharged. Both patient and endoscopist satisfaction will be measured on a scale of 0 to 5 using Likert scale. This comprehensive approach aims to determine the efficacy, safety, and patient/endoscopist experience associated with the three sedative regimens during colonoscopy

ELIGIBILITY:
Inclusion criteria:

* Adults aged 18-60 years
* Both Genders
* Indication of colonoscopy procedure without advanced intervention
* American Society of Anesthesiologists (ASA) physical status I or II
* Competent to give informed consent
* Exclusion criteria:
* Personal history of allergic reaction or other contra-indications to midazolam, propofol or fentanyl
* Age below 18 or above 60 years
* Chronic use of benzodiazepines
* ASA physical status III or above
* Pregnancy
* History of smoking or alcohol abuse
* Body mass index > 35 kg/m2
* History of airway obstruction or difficult intubation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 157 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Degree of sedation | every 3 minutes till the end of procedure
  The degree of sedation shows the depth of sedation. It will be measured by the Observer's assessment of alertness/sedation scale with a minimum and maximum value of 1 and 5 reflecting depth of sedation. Where score 1 means deeply sedated while score 5 means fully awake. Higher scores means not enough sedation.
Onset of sedation | It will be measured every 1 minute till 20 minutes.
  Onset of sedation means how rapidly patient is sedated after giving the sedative medication. if after 20 minutes, patient not sedated then it will be considered failed to sedate.
Adverse events and complication | Monitored continuously during procedure and post procedure for 2 hours and then up to 48 hours after discharge on telephone
  Adverse events are any unintended or undesirable clinical occurrences that arise during or after a medical procedure, treatment, or intervention. These events may be related to the procedure itself, the medications administered. These may include hypotension, bradycardia, tachycardia, hypoxia, oversedation leading to respiratory suppression

SECONDARY OUTCOMES:
Patient's satisfaction with the procedure | 2 hours from the start of the procedure.
  It reflects patient's overall satisfaction about the colonoscopy procedure under given sedation. It will be assessed on Likert scale with minimum and maximum values of 1 to 5. On the Linkert scale 5 is maximum satisfaction and 1 is the least.
procedure completion rate | Decision for procedure completion successfully or not will be at 1 hour. Procedure completion rate at 6 months
  The colonoscopy procedure will be considered successful if the endoscopist examines the colon from the rectum to the cecum. it will be done at 1 hour.The procedure completion rate, representing the percentage of successful procedures, will be calculated six months after collecting all data from the study.

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud Hospital, Unaizah, Al-Qassim Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
IPD data will not be shared

DOCUMENTS (1):
  • Study Protocol (2025-01-06): https://cdn.clinicaltrials.gov/large-docs/05/NCT06763705/Prot_000.pdf